CLINICAL TRIAL: NCT06448156
Title: Epidemiological Study of Out-of-hospital Cardiac Arrest in Guangzhou
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: MR-44-24-003181
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Arrest; Sudden Cardiac Death
MeSH Terms: conditions — Heart Arrest; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- 0-19 years age group
  Interventions: Diagnostic Test: "cardiac arrest" and "sudden death"
- 20-29 years age group
  Interventions: Diagnostic Test: "cardiac arrest" and "sudden death"
- 30-39 years age group
  Interventions: Diagnostic Test: "cardiac arrest" and "sudden death"
- 40 to 49 age group
  Interventions: Diagnostic Test: "cardiac arrest" and "sudden death"
- 50 to 59 age group
  Interventions: Diagnostic Test: "cardiac arrest" and "sudden death"
- 60 to 69 age group
  Interventions: Diagnostic Test: "cardiac arrest" and "sudden death"
- 70 to 79 age group
  Interventions: Diagnostic Test: "cardiac arrest" and "sudden death"
- 80+age group: Age group greater than or equal to 80 years
  Interventions: Diagnostic Test: "cardiac arrest" and "sudden death"

INTERVENTIONS:
Diagnostic Test: "cardiac arrest" and "sudden death" — Selection of cases with a secondary diagnosis containing the diagnostic keywords "cardiac arrest" and "sudden death"."cardiac arrest" and "sudden death".The incidence rate is then calculated

SUMMARY:
Aim This was a population-based retrospective cohort study of OHCA. This study intends to retrospectively analyze the data of pre-hospital emergency system in Guangzhou for 10 years, explore the incidence trend of OHCA in Guangzhou for 10 years; Through further analysis, we try to explore the time distribution characteristics of OHCA in order to understand the epidemiological characteristics and rules of OHCA in super large cities in southern China.

Methods The pre-hospital traffic data in the main urban area of Guangzhou Emergency Medical Command Center database from 2011 to 2020 were collected. The cases diagnosed as "cardiac arrest" and "sudden death" were screened, and the cases with non-cardiac causes in the diagnosis were deleted. The crude incidence rate and age-standardized incidence rate of OHCA were calculated. Joinpoint software was used to calculate the changing nodes in the OHCA incidence trend, and the AnnualPercent Change (APC) and Average AnnualPercent Change (Average AnnualPercent Change, APC) of OHCA incidence were calculated. AAPC). The OHCA data were grouped according to the six main urban areas, and the crude incidence rate, ASIR and changing trend of the six main urban areas were calculated. The data of OHCA were grouped by age, and the crude incidence rate, ASIR and changing trend of each age group were calculated. The data information was divided into groups according to 24 hours a day, 7 days a week, and four seasons. The number of OHCA cases in different time periods was statistically described. The data were imported into SPSS 26.0 for analysis, and Mann-Kendall test was used to evaluate the statistical significance of the time trend. Time rhythm variability was tested for mean distribution using chi-square goodness of fit test.

ELIGIBILITY:
Inclusion Criteria:

Cases in the database with a secondary diagnosis containing the diagnostic keywords "cardiac arrest" and "sudden death"

Exclusion Criteria:

1. cases where the diagnosis of "cardiac arrest" and "sudden death" includes a diagnosis of a non-cardiac cause such as asphyxiation, suicide, drowning, advanced cancer, trauma, shock, poisoning, cerebral vascular accident, etc;
2. cases with duplicate records of sex, age, time of call, pick-up address and initial diagnosis

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases in the database with a secondary diagnosis containing the diagnostic keywords "cardiac arrest" and "sudden death".Data were collected from the GZ-EMS Command Centre's dispatch system database of pre-hospital data for the central urban districts of City.
Sampling Method: Non-Probability Sample
Enrollment: 44375 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Crude incidence rate | 2011-01-01 to 2020-12-31
  The frequency of new cases of a disease in a given population over a given period of time.
Age standardized incidence rate | 2011-01-01 to 2020-12-31
  Incidence rates after removing the influence of age, and incidence rates normalised by age. The rationale is that age is an important influence on cancer incidence, with higher incidence rates occurring at older ages, so that if the age structure of the population in two regions is very different, it is not possible to determine whether the high incidence of a disease in a particular region is due to a different age composition or to other influences if incidence rate comparisons are applied.
Average annual percentage change | 2011-01-01 to 2020-12-31
  Calculated using the weighted average of the APC, it is an overall measure of trend.
Annual percentage change | 2011-01-01 to 2020-12-31
  Indicates the change from one year to the next within a segment at a constant percentage on a log-linear model for evaluating trends within segments.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Yu, Study Director — Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, China
Locations (1):
- Yu Tao, Guangdong, Guangdong, China

IPD SHARING:
Plan to Share IPD: No